CLINICAL TRIAL: NCT00860821
Title: A Randomised, Double-blind, Placebo-controlled, Two-way Crossover, Single-centre Methodologhy Study in Healthy Subjects to Evaluate the Effect of Oral Dosing With AZD8309 on Cells and Inflammatory Biomarkers in Nasal Lavage and Blood After Nasal Challenge With Lipopolysaccharide (LPS).
Brief Title: A Methodology Study in Healthy Subjects to Evaluate the Effect of AZD8309 After Nasal Administration of Lipopolysaccharide (LPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Leif Eriksson, MD PhD, Medical Science Director, RITA CPT2, AstraZeneca R&D Lund
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1511M00004
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Healthy subjects; LPS; Effect; Intranasally
MeSH Terms: interventions — AZD8309

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD8309
  Interventions: Drug: AZD8309
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: AZD8309

INTERVENTIONS:
Drug: AZD8309 — oral solution 30 mg/g, dose: 300mg bid for 3 days
  Arms: 1
Drug: AZD8309 — oral solution 30 mg/g, dose: 300mg bid for 3 days
  Arms: 2

SUMMARY:
The purpose of this methodology study is to evaluate the effect of AZD8309 on cells and inflammatory biomarkers in nasal lavage and blood after nasal challenge with lipopolysaccharide (LPS)

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or healthy, permanently sterilized, women aged 18 to 50 years inclusive, non-smokers or ex-smokers, Body Mass Index 18 to 30 kg/m2 and minimum body weight of 50 kg
* Blood neutrophil count above 2.2x10^9/L

Exclusion Criteria:

* Clinical relevant disease and/or abnormality

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Neutrophil numbers in nasal lavage | 3 times each in the end of two treatment periods

SECONDARY OUTCOMES:
Cells and inflammatory biomarkers in nasal lavage | 3 times in the end of the two treatment periods
Cells and inflammatory biomarkers in blood | 2 times in the beginning and 5 times in the end of the two treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Lars Olaf Cardell, Principal Investigator — Department of Otorhinolaryngology, Malmö University Hospital, Sweden; Leif Eriksson, Study Director — AstraZeneca R&D Lund, Sweden
Locations (1):
- Research Site, Malmo, Sweden

REFERENCES:
- [Derived] Leaker BR, Barnes PJ, O'Connor B. Inhibition of LPS-induced airway neutrophilic inflammation in healthy volunteers with an oral CXCR2 antagonist. Respir Res. 2013 Dec 16;14(1):137. doi: 10.1186/1465-9921-14-137. PMID 24341382